CLINICAL TRIAL: NCT02804490
Title: Efficacy of Biofortified Maize to Improve Maternal and Infant Vitamin A Status
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: University of California, Davis (Other); Newcastle University (Other); HarvestPlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014H8314.JHU
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Vitamin A Deficiency
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- White maize (Placebo Comparator): Conventional maize flour
  Interventions: Dietary Supplement: Conventional white maize
- Biofortified maize (Experimental): Provitamin A carotenoid biofortified maize flour
  Interventions: Dietary Supplement: Provitamin A carotenoid biofortified maize
- Fortified maize (Active Comparator): Retinyl palmitate fortified maize flour
  Interventions: Dietary Supplement: Preformed vitamin A fortified maize

INTERVENTIONS:
Dietary Supplement: Conventional white maize — Women and their infants will receive 2 meals/day prepared with conventional white maize flour (287 g dry weight/d for women; 50 g dry weight/d for infants), 6 days/week for 15 weeks
  Arms: White maize
Dietary Supplement: Provitamin A carotenoid biofortified maize — Women and their infants will receive 2 meals/day prepared with provitamin A carotenoid biofortified orange maize flour (287 g dry weight/d for women; 50 g dry weight/d for infants), 6 days/week for 15 weeks
  Arms: Biofortified maize
Dietary Supplement: Preformed vitamin A fortified maize — Women and their infants will receive 2 meals/day prepared with preformed vitamin A fortified, conventional white maize flour (287 g dry weight/d for women; 50 g dry weight/d for infants), 6 days/week for 15 weeks
  Arms: Fortified maize

SUMMARY:
The purpose of this randomized control trial is to test the impact of provitamin A carotenoid biofortified maize meal consumption on maternal and infant vitamin A status.

DETAILED DESCRIPTION:
Vitamin A deficiency remains a major public health problem in low and middle income countries. Approximately 50% of Zambian children are thought to be affected. This randomized control trial will test the efficacy of provitamin A carotenoid biofortified maize meal consumption as a strategy to improve vitamin A status among lactating Zambian mothers and their infants. The investigators will enroll up to 255 mother/infant pairs to a three-month study, during which they will receive one of the following three interventions: 1) conventional white maize, 2) provitamin A carotenoid biofortified orange maize, or 3) preformed vitamin A fortified white maize.

ELIGIBILITY:
Inclusion Criteria:

* Singleton birth
* No birth defects
* Free from chronic health conditions
* Infant received 100,000 IU vitamin A at 6 months of age
* Currently breastfeeding
* Not pregnant at 9 months post partum
* Hemoglobin > 8.0 g/dL for women and > 7.0 g/dL for infants

Exclusion Criteria:

* Multiple birth
* Birth defects
* Any chronic health condition requiring regular medical visits
* Infant did not receive vitamin A capsule at 6 months of age
* No longer breastfeeding
* Pregnant
* Hemoglobin ≤ 8.0 g/dL for women or ≤ 7.0 g/dL for infants

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Infant vitamin A stores | 90 days
  Total body vitamin A stores of infants measured by retinol isotope dilution

SECONDARY OUTCOMES:
Maternal breast milk retinol | 90 days
  Breast milk retinol concentrations of women measured by high performance liquid chromatography
Maternal plasma retinol | 90 days
  Plasma retinol concentrations of women measured by high performance liquid chromatography
Maternal dark adaptation | 90 days
  Pupillary responsiveness of women measured by portable field dark adaptometer

CONTACTS AND LOCATIONS:
Overall Officials: Amanda C Palmer, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Marjorie Haskell, PhD, Study Director — University of California, Davis; Rose Mwanza, MD, Study Director — Provincial Medical Office, Central Province, Zambia
Locations (1):
- JHU Office, Mkushi, Central Province, Zambia

REFERENCES:
- [Background] Gannon B, Kaliwile C, Arscott SA, Schmaelzle S, Chileshe J, Kalungwana N, Mosonda M, Pixley K, Masi C, Tanumihardjo SA. Biofortified orange maize is as efficacious as a vitamin A supplement in Zambian children even in the presence of high liver reserves of vitamin A: a community-based, randomized placebo-controlled trial. Am J Clin Nutr. 2014 Dec;100(6):1541-50. doi: 10.3945/ajcn.114.087379. Epub 2014 Oct 8. PMID 25411289
- [Background] Palmer AC, Siamusantu W, Chileshe J, Schulze KJ, Barffour M, Craft NE, Molobeka N, Kalungwana N, Arguello MA, Mitra M, Caswell B, Klemm RD, West KP Jr. Provitamin A-biofortified maize increases serum beta-carotene, but not retinol, in marginally nourished children: a cluster-randomized trial in rural Zambia. Am J Clin Nutr. 2016 Jul;104(1):181-90. doi: 10.3945/ajcn.116.132571. Epub 2016 May 11. PMID 27169838
- [Background] Oxley A, Berry P, Taylor GA, Cowell J, Hall MJ, Hesketh J, Lietz G, Boddy AV. An LC/MS/MS method for stable isotope dilution studies of beta-carotene bioavailability, bioconversion, and vitamin A status in humans. J Lipid Res. 2014 Feb;55(2):319-28. doi: 10.1194/jlr.D040204. Epub 2013 Oct 24. PMID 24158962
- [Background] Labrique AB, Palmer AC, Healy K, Mehra S, Sauer TC, West KP Jr, Sommer A. A novel device for assessing dark adaptation in field settings. BMC Ophthalmol. 2015 Jul 9;15:74. doi: 10.1186/s12886-015-0062-7. PMID 26156587
- [Background] Muzhingi T, Gadaga TH, Siwela AH, Grusak MA, Russell RM, Tang G. Yellow maize with high beta-carotene is an effective source of vitamin A in healthy Zimbabwean men. Am J Clin Nutr. 2011 Aug;94(2):510-9. doi: 10.3945/ajcn.110.006486. Epub 2011 Jun 29. PMID 21715509
- [Background] Li S, Nugroho A, Rocheford T, White WS. Vitamin A equivalence of the ss-carotene in ss-carotene-biofortified maize porridge consumed by women. Am J Clin Nutr. 2010 Nov;92(5):1105-12. doi: 10.3945/ajcn.2010.29802. Epub 2010 Sep 1. PMID 20810977
- [Derived] Palmer AC, Jobarteh ML, Chipili M, Greene MD, Oxley A, Lietz G, Mwanza R, Haskell MJ. Biofortified and fortified maize consumption reduces prevalence of low milk retinol, but does not increase vitamin A stores of breastfeeding Zambian infants with adequate reserves: a randomized controlled trial. Am J Clin Nutr. 2021 May 8;113(5):1209-1220. doi: 10.1093/ajcn/nqaa429. PMID 33693468